CLINICAL TRIAL: NCT00003614
Title: Phase II Study of Weekly Paclitaxel by 1-HR Infusion Plus Estramustine in Metastatic Hormone-Refractory Prostate Carcinoma
Brief Title: Paclitaxel Plus Estramustine in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066691; E-1898
Record Dates: First submitted 2000-11-06; First posted 2004-05-24 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; Paclitaxel

INTERVENTIONS:
Drug: estramustine phosphate sodium
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel plus estramustine in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of weekly paclitaxel plus estramustine on PSA response in patients with metastatic hormone-refractory prostate cancer. II. Describe the toxic effects of this treatment in this patient population. III. Determine the effect of treatment on pain, asthenia, and quality of life. IV. Determine the objective response rate after treatment among the patients with bidimensionally measurable disease.

OUTLINE: Patients receive estramustine orally twice a day on days 1-3 of each week for 6 weeks. Patients also receive paclitaxel IV over 1 hour on day 2 of each week for 6 weeks. Courses repeat every 8 weeks in the absence of unacceptable toxicity and disease progression. Quality of life is assessed prior to treatment and at weeks 4, 8, 20, and 24. Patients are followed every 3 months for 2 years, every 6 months for years 2-5, and then annually thereafter.

PROJECTED ACCRUAL: There will be 17-52 patients accrued into this study over 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic hormone-refractory adenocarcinoma of the prostate gland Elevated serum acid phosphatase or PSA levels must not be only evidence of disease Must have evidence of progressive metastatic disease (e.g., bone, pelvic mass, lymph node, liver, or lung metastases) Radiological evidence of hydronephrosis alone does not constitute evidence of metastatic disease Patients with bone metastases only (i.e., lacking measurable soft tissue disease) must have PSA level of at least 20 ng/mL Patients with soft tissue metastases and/or visceral disease must have either bidimensionally measurable disease or a PSA level of at least 20 ng/mL Must have had prior treatment with bilateral orchiectomy or other primary hormonal therapy (e.g., estrogen therapy, LHRH-blocker plus flutamide, etc.) with evidence of treatment failure No carcinomatous meningitis or brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 OR Granulocyte count at least 2,000/mm3 Platelet count greater than 100,000/mm3 No history of deep venous thrombosis Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT and SGPT no greater than 2 times normal Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: No active angina pectoris No known New York Heart Association class II-IV heart disease No history of myocardial infarction in the last 6 months Other: No history of prior malignancy except if curatively treated and disease free for time period considered appropriate for cure of specific cancer No other serious concurrent illness or active infection Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy (including neoadjuvant chemotherapy) Endocrine therapy: See Disease Characteristics At least 6 weeks since prior bicalutamide At least 4 weeks since prior flutamide or nilutamide Recovered from prior toxicities of endocrine therapy Radiotherapy: No prior strontium 89, samarium 153, or other radioisotope therapies At least 4 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics Recovered from prior surgery

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02-04 (Actual); Primary Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Hudes, MD, Study Chair — Fox Chase Cancer Center
Locations (28):
- United States (27):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Hospitals, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Hudes GR, Manola J, Conroy J, et al.: Phase II study of weekly paclitaxel (P) by 1-hour infusion plus reduced-dose oral estramustine (EMP) in metastatic hormone-refractory prostate carcinoma (HRPC): a trial of the Eastern Cooperative Oncology Group. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-697, 2001.